CLINICAL TRIAL: NCT01089634
Title: Left Ventricular Capture Management (LEARN) Study
Brief Title: Left Ventricular Capture Management Study
Acronym: LEARN
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: LEARN2007
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia; Bradyarrhythmia
Keywords: LV measurement; CRT; Concerto; LVCM; LV threshold; new CRT
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Bradycardia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objective:

To characterize left ventricular (LV) threshold behavior over time using daily left ventricular capture management (LVCM) measurements.

Study Design:

This is a multicenter, prospective, non-interventional study with patients receiving their first cardiac resynchronisation therapy-implantable cardioverter defibrillator (CRT-ICD) device. The study design, based on the primary objective, is an observational examination of LV thresholds over time. Daily left ventricular threshold measurements will be collected using the LVCM feature. Up to 150 patients will be enrolled in Canada to evaluate the primary objective at up to 15 study centers.

Data will be collected at Baseline, Implant, 12 months post-implant and all regularly scheduled follow-up visits up to 12 months post-implant.

Devices:

The ConcertoTM CRT-ICD device and future Medtronic CRT-ICD devices containing the LVCM feature will be used in this study.

DETAILED DESCRIPTION:
I. Study Purpose:

The purpose of the LEARN Study is to provide information that will assist clinicians in managing LV thresholds.

II. Device Description:

The CRT-ICD devices to be used in this study are all Therapeutic Products Directorate licensed, market released Medtronic CRT-ICD devices equipped with the LVCM feature. Currently this includes only the ConcertoTM CRT Defibrillator. Future Medtronic models equipped with the LVCM feature that become Therapeutic Products Directorate licensed and market released in the future are also included.

The study will allow all commercially available leads from all manufacturers that are compatible with Medtronic CRT-ICD devices. Devices will be programmed and interrogated with a Medtronic 9790 or 2090 programmer.

Medtronic defibrillators automatically detect and treat episodes of ventricular fibrillation (VF), ventricular tachycardia (VT) and bradyarrhythmia. When a ventricular arrhythmia is detected, the implantable devices deliver defibrillation, cardioversion, anti-tachycardia pacing or standard pacing therapy to terminate the ventricular arrhythmia. In addition, Medtronic CRT defibrillators, including Concerto, also provide Cardiac Resynchronization therapy. All devices in this study will be used according to their intended use.

III. Study Objective:

Primary Study Objective: To characterize LV threshold behavior over time.

IV. Study Scope:

150 patients will be enrolled in Canada to evaluate the primary objective at up to 15 study centers. Individual centers will be limited to a maximum of 30 enrollments.

Patients will be followed for a 12 month period with interim visits occurring according to regular clinic follow up schedules.

V. Methodology:

A. Study Design This is a multicenter, prospective, non-interventional study with patients receiving their first CRT-ICD device. The study design, based on the primary objective, is an observational examination of LV thresholds.

Patients will be followed in clinic as per the hospital ICD clinic standard follow up schedule with a mandatory follow-up visit at 12 months (± 30 days) post-implant. The following will be collected at the 12 month (± 30 days) visit and at all regularly scheduled follow-up visits: LV threshold measurements, changes in cardiovascular medications and a save to disk file.

B. Patient Population Inclusion Criteria

* Patients who will be implanted with their first CRT defibrillator system.
* Patients who will be implanted with a Medtronic CRT defibrillator containing the LVCM feature.
* Patients who are willing and able to sign an IRB/MEC approved patient informed consent.
* Patients who are geographically stable and available for follow-up at the study center for the required follow-up duration of the study

Exclusion Criteria

Patients who meet any of the following criteria are excluded from entry into the study:

* Patients who have a pre-existing LV lead prior to enrollment
* Patients who have a life expectancy of less than 1 year
* Patients included in another clinical trial that will affect the objectives of this study

VI. Study Procedures:

A. Overview of Data Collection Requirements:

Clinical data will be collected at baseline, implant, regularly scheduled follow-up visits over 12months, system modifications, and patient withdrawal/exit.

Data will be collected via case report forms, and Save-to-Disk files.

B. Enrollment Procedures:

There are no medications or treatments that are required in this study. Patients enrolled in the LEARN Study will receive the standard of medical care that is typically provided by the investigator. There are no medications or treatments that are not permitted in this study, unless they conflict with the patient inclusion/exclusion criteria.

Patients planned to be implanted with a CRT-ICD will be evaluated for inclusion and exclusion criteria. Patients who meet these inclusion and exclusion criteria will be invited to participate in the study. Each study subject must sign an IRB/MEC approved consent form prior to implant. Once the patient signs the consent form the patient is enrolled in the LEARN Study. Patients must be consented and enrolled prior to hospital discharge.

At the time of enrollment, a Baseline Case Report Form must be completed. The following information will be documented on this form:

* Verification that all inclusion/exclusion criteria were met
* Patient demographic information
* Cardiovascular status and history
* Arrhythmia status and history
* Current Cardiovascular and Medications

C. Implant Procedures:

The Medtronic device will be implanted according to the manufacturer's instructions. The leads will be implanted according to the instructions provided with the applicable lead. Only commercially available RA, RV and LV leads may be used in this study.

At implant, record the model number and serial number of the device and leads implanted on the implant form.

In the event that a patient does not receive a ConcertoTM or equivalent LVCM equipped Medtronic CRT-ICD device, they will be withdrawn from the study via a study exit case report form. In the event that an LV lead cannot be placed at the time of implant and subsequent attempts to implant an LV lead are either not successful or not attempted, the patient will be withdrawn from the study via a study exit case report form.

D. LVCM Programming Requirements:

In order to collect data on LV thresholds, the LVCM feature must be set to either Monitor or Adaptive. The setting must be noted on the implant form.

E. Follow-up Procedures:

The following will be performed at all regularly scheduled in-clinic follow-up visits for 12 months post-implant including the required 12 month visit. Record the required data on the corresponding CRF for each patient.

1. Record LV lead data on the follow up CRF.
2. Record results of manual LV threshold testing

b) 'Interrogate all' and perform a final Save-to-Disk.

F. Adverse Event Reporting:

Adverse events will not be collected in this study.

G. System Modification:

In the event that the CRT defibrillator or lead system requires invasive modification (e.g., device or LV lead explant, device or LV lead replacement, attempting to place LV lead after initial failed attempt, or lead repositioning), the System Modification Case Report Form must be completed.

If the patient's CRT defibrillator system or LV lead is explanted and not replaced, complete a study exit form and exit the patient from the study.

H. Study Exit:

In the event that a patient is unable or unwilling to continue participation in the study, notify the Medtronic Clinical Research Manager immediately.

Patients who are enrolled in the study, but do not receive a Concerto or equivalent Medtronic device, as well as patients who do not receive an LV lead must be withdrawn via a Study Exit Case Report Form.

If a patient expresses desire to withdraw from the study, a Study Exit Case Report Form must be completed. The reason for patient withdrawal must be documented on this form.

In the case that the patient fails to comply with the follow-up schedule, the study site must attempt to contact the patient. Each attempt to contact the patient must be documented in the patient's records. In the event that the patient is lost to follow-up, a Study Exit Case Report Form must be completed. Details on all attempts to contact the patient and the method used (e.g. telephone, registered mail) must be recorded on the case report form.

In the event of a patient death, a study exit form should be completed with patient death listed as the reason for withdrawal.

I. Study Deviations:

A Study Deviation is defined as an event where the clinical Investigator or site personnel did not conduct the study according to the Investigational Plan, protocol, applicable laws or regulations or the Investigator Agreement. Examples include but are not limited to: failure to obtain informed consent, missing save to disk etc. It is the responsibility of the investigator to notify the study sponsor (Medtronic of Canada Ltd.) of any deviation and complete the Deviation CRF including rationale for the deviation. Any planned deviation that may affect the rights, safety or welfare of a patient involved in this study requires prior approval of the IRB/MEC and Medtronic. If a patient is enrolled in violation of the inclusion and exclusion criteria, the patient will not contribute to the study objectives. All protocol deviations should be reported by the investigator to Medtronic on a deviation CRF and to the sites IRB/MEC as per IRB/MEC policy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be implanted with their first CRT defibrillator system.
* Patients who will be implanted with a Medtronic CRT defibrillator containing the LVCM feature.
* Patients who are willing and able to sign an IRB/MEC approved patient informed consent.
* Patients who are geographically stable and available for follow-up at the study center for the required follow-up duration of the study

Exclusion Criteria:

* Patients who have a pre-existing LV lead prior to enrollment
* Patients who have a life expectancy of less than 1 year
* Patients included in another clinical trial that will affect the objectives of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients who will be implanted with their first CRT defibrillator system.
  * Patients who will be implanted with a Medtronic CRT defibrillator containing the LVCM feature.
  * Patients who are willing and able to sign an IRB/MEC approved patient informed consent.
  * Patients who are geographically stable and available for follow-up at the study center for the required follow-up duration of the study
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2007-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McCann, R.N., MBA, Study Chair — Medtronic; Allison Rubino, Study Chair — Medtronic
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada